CLINICAL TRIAL: NCT01632137
Title: A Phase 3 Study to Determine the Efficacy and Safety of Rebamipide in Subjects With Dry Eye Syndrome
Brief Title: Efficacy and Safety of Rebamipide in Subjects With Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU-RED-301
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo (vehicle)
- Rebamipide 2% ophthalmic suspension (Experimental)
  Interventions: Drug: Rebamipide 2% ophthalmic suspension

INTERVENTIONS:
Drug: Rebamipide 2% ophthalmic suspension — Instill one drop into each eye 4 times a day for 4 weeks.
  Arms: Rebamipide 2% ophthalmic suspension
Drug: Placebo (vehicle) — Instill one drop into each eye 4 times a day for 4 weeks.
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rebamipide ophthalmic suspension in subjects with dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* History of dry eye-related ocular symptoms for at least 20 months.
* Meet protocol-defined criteria for corneal and conjunctival staining.
* Meet protocol-defined criteria for ocular discomfort.

Exclusion Criteria:

* Active anterior segment ocular disease other than dry eye syndrome.
* Inability to suspend the use of topical ophthalmic medications throughout the duration of the study.
* Inability to suspend the use of contact lenses for the duration of the study.
* Judged by the investigator to be ineligible for the study because of a past or concurrent systemic disease, or safety concerns.
* Received any other investigational product within 4 months before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Primary ocular sign: Fluorescein corneal staining total score | 4 weeks
Primary ocular symptom: Worst ocular symptom severity score | 4 weeks

SECONDARY OUTCOMES:
Fluorescein corneal staining total score | 2 weeks
Worst ocular symptom severity score | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Acucela Medical Monitor, Study Director — Kubota Vision Inc.
Locations (34):
- United States (34):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Artesia, California
  - Glendale, California
  - Inglewood, California
  - San Diego, California
  - Wheat Ridge, Colorado
  - Fort Myers, Florida
  - Miami, Florida
  - Plantation, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Morrow, Georgia
  - Baton Rouge, Louisiana
  - Lutherville, Maryland
  - Kansas City, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Las Vegas, Nevada
  - Princeton, New Jersey
  - Rochester, New York
  - Rockville Centre, New York
  - Valley Stream, New York
  - Wantagh, New York
  - Ashville, North Carolina
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Mason, Ohio
  - Pittsburgh, Pennsylvania
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia